CLINICAL TRIAL: NCT06383260
Title: Assessing the Prevalence of Attention Deficit Hyperactivity Disorder (ADHD) Symptoms in Undiagnosed Young Adults:A Cross Sectional Study
Status: Completed | Type: Observational
Sponsor: Jinnah Sindh Medical University (Other)
Responsible Party: Principal Investigator, Aina Marzia Syed, Aina Marzia Syed, Jinnah Sindh Medical University
Other Study IDs: 009-0001-7719-1189
Record Dates: First submitted 2024-04-21; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Finding the Prevalence of ADHD in Undiagnosed Young Adults

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Age group: 18-20 21-22 22-24
- ASRS V1.1 scores(%): Score of Ahdh self report scale questionnaire
  Interventions: Behavioral: Behavioral diagnostic
- ADHD symptom prevalence: People who got more than 4 in part A of questionnaire and more than 6 in Part B
  Interventions: Behavioral: Behavioral diagnostic

INTERVENTIONS:
Behavioral: Behavioral diagnostic — Diagnosing the behavioral pattern
  Groups: ADHD symptom prevalence; ASRS V1.1 scores(%)

SUMMARY:
To asses the prevalence of Attention deficit hyperactivity disrorder in undiagnosed young adults.

DETAILED DESCRIPTION:
Finding the prevalence of Attention Deficit Hyperactivity Disorder (ADHD) in undiagnosed young adults using the questionnaire provided by WHO ,

ELIGIBILITY:
Inclusion Criteria:

* undiagnosed

Exclusion Criteria:

* diagnosed with any mental disability

Ages: 18 Years to 24 Years | Sex: All
Age Groups: Adult
Study Population: Young adults between age group of 18-24
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Assess the prevalence of undiagnosed ADHD in Young adults | 2 months
  To find out the prevalence of ADHD in Young adults

CONTACTS AND LOCATIONS:
Overall Officials: Aina M Syed, Principal Investigator — Jinnah Sindh Medical University
Locations (1):
- JSMU, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT06383260/Prot_SAP_000.pdf